CLINICAL TRIAL: NCT00146588
Title: A Pilot Study of Cytoxan, Epirubicin, and Capecitabine in Women With Stage I/II/IIIA Breast Cancer
Brief Title: Cytoxan, Epirubicin and Capecitabine in Women With Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Craig A. Bunnell, MD, MPH (Other)
Collaborators: Dana-Farber Cancer Institute (Other); Massachusetts General Hospital (Other); Brigham and Women's Hospital (Other); Beth Israel Deaconess Medical Center (Other); Pharmacia (Industry)
Responsible Party: Sponsor-Investigator, Craig A. Bunnell, MD, MPH, Associate Chief Medical Officer, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 02-036
Record Dates: First submitted 2005-09-06; First posted 2005-09-07 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2014-10

CONDITIONS: Breast Cancer; Stage I Breast Cancer; Stage II Breast Cancer; Stage IIIA Breast Cancer
Keywords: Breast cancer; cytoxan; epirubicin; capecitabine
MeSH Terms: conditions — Breast Neoplasms | interventions — Cyclophosphamide; Epirubicin; Capecitabine

INTERVENTIONS:
Drug: Cyclophosphamide — Intravenously on day 1 of each 21-day treatment cycle for 12-18 weeks depending upon response.
  Other Names: Cytoxan
Drug: Epirubicin — Intravenously on day 1 of each 21-day treatment cycle for 12-18 weeks depending upon response.
Drug: Capecitabine — Given orally on days 4-17 of each 21-day treatment cycle for 12-18 weeks depending upon response.

SUMMARY:
The purpose of this study is to find out what effects (good and bad) a combination of cytoxan, epirubicin, and capecitabine have on women with Stage II/II/IIIA breast cancer.

DETAILED DESCRIPTION:
* Each treatment cycle lasts 21 days and patients will participate in a least 4 cycles, but no more than 6 cycles of treatment.
* Patients will receive cytoxan (cyclophosphamide) and epirubicin intravenously on day 1 of each treatment cycle. On days 4-17 of each cycle, patients will take capecitabine orally twice a day.
* While on the study patients will be required to complete a diary of they capecitabine treatment.
* Blood tests will be performed each week along with surveys at the beginning of the trial and certain follow-up visits to evaluate the patient's experience with the oral chemotherapy.
* Patients will be on the treatment for 12-18 weeks depending upon whether or not the disease progresses or the patient develops inacceptable side effects.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed Stage I-III breast cancer. If Stage I, should be deemed of sufficiently high risk of developing recurrent disease to warrant participation.
* 18 years of age or older
* ANC > 1,000/mm3
* Platelet count > 100,000/mm3
* Hemoglobin > 10
* Creatinine < 2.0
* SGOT < 2 x ULN
* Bilirubin < 1.5mg/dl
* Able to swallow and retain oral medication
* LVEF greater than or equal to 50%
* ECOG performance status of 0 or 1

Exclusion Criteria:

* Pregnant or lactating
* Prior malignancy within 5 years (excluding squamous or basal cell skin cancers)
* Prior chemotherapy within 5 years
* Prior anthracycline therapy
* Serious comorbid physical or psychological condition

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2002-04; Primary Completion 2004-12 (Actual); Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
To determine the feasibility of administering cytoxan, epirubicin, and capecitabine to women with Stage I/II/IIIA breast cancer. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Craig Bunnell, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Center, Boston, Massachusetts